CLINICAL TRIAL: NCT05845632
Title: Association Between Time to Treatment and Disease-free Survival of Patients With High-risk Cutaneous Squamous Cell Carcinoma in the Head and Neck Region.
Brief Title: Time to Treatment and Disease-free Survival of Patients With High-risk Head-neck Cutaneous Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-2885-A-2
Record Dates: First submitted 2023-04-17; First posted 2023-05-06 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Carcinoma, Squamous Cell; Skin Cancer; Carcinoma, Squamous Cell, Skin; Carcinoma, Squamous Cell of Head and Neck; Recurrence; Metastasis
Keywords: Disease free survival; Survival; Multicenter; Time to treatment; Waiting times
MeSH Terms: conditions — Carcinoma, Squamous Cell; Skin Neoplasms; Carcinoma; Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Short time to treatment (<30 days): Patients with high-risk HNcSCC with a time to treatment (date of pathological diagnosis to date of start treatment) of less than 30 days.
  Interventions: Other: Treatment
- Long time to treatment (30 days or more): Patients with high-risk HNcSCC with a time to treatment (date of pathological diagnosis to date of start treatment) of 30 days or more.
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — Patients were treated with surgery, radiotherapy or surgery with postoperative radiotherapy.

SUMMARY:
The purpose of this study is to investigate the association between time to treatment (defined as date of pathological diagnosis to date of start treatment) and disease free survival in patients with high risk cutaneous squamous cell carcinoma in the head-neck region.

DETAILED DESCRIPTION:
Skin cancer is the most common type of cancer in the Netherlands. Cutaneous squamous cell carcinoma (cSCC) accounts for 20% of all cutaneous malignancies. The incidence of cSCC has been rising over the years in the Netherlands, from 8,966 new cSCCs cases registered in 2012 to 14,873 cases in 2022. cSCCs mostly involve patients aged 75 years and older. Since exposure to UV radiation is the main risk factor for the development, cSCCs particularly occur on sun exposed areas of the skin such as in the head-neck region and the extremities. Other risk factors include a Fitzpatrick skin type I or II, use of immunosuppression, exposure to arsenic, and infection with human papilloma virus.

Risk of metastasis and recurrence in general cSCCs are 2.6-5% and 1.9-3.7%, respectively. However, these risk ratios may increase to 37% in high-risk cSCCs. High risk cSCCs are defined as cSCCs with risk factors for development of metastatic disease or recurrence, e.g. poor histological differentiation, perineural/lymphovascular infiltration, diameter ≥20 mm.

Due to the increasing incidence, advanced age, risk of metastasis and recurrence, and the high risk-location in the head-neck region related to functional and cosmetic importance, high-risk cSCCs in the head-neck region (high-risk HNcSCCs) require complex and multidisciplinary care. Therefore, care pathways have been developed. An important part of these care pathways are waiting times and, in particular, the time to treatment. For example, in mucosal head-neck tumors, prolonged waiting times have been described to be associated with reduced survival rates. This led to the hypothesis that prolonged waiting times result result in lower survival rates for patients with high-risk HNcSCCs. This study aimed to investigate the association between time to treatment defined as date of pathological diagnosis to date of start treatment) and disease free survival in patients with high risk HNcSCCs.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with high-risk HNcSCCs, defined as T2 to T4 HNcSCC
* Treated in the Maastricht University Medical Center+ (MUMC+) or Radboud University Medical Center (RadboudUMC)
* Treated between 2010 to 2018

Exclusion Criteria:

* Patients aged younger than 18 years
* Patients with a T1 HNcSCC
* Patients with recurrence or metastatic disease of a previously treated HNcSCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathology reports of patients, aged 18 years or older, diagnosed with a T2 to T4 high-risk HNcSCC, treated in the MUMC+ or Radboud UMC between 2010 and 2018, will be obtained from the Pathological Anatomical National Automated Archive (PALGA).
Sampling Method: Non-Probability Sample
Enrollment: 965 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Association time to treatment and survival | 5 years after treatment
  The association between time to treatment (in days) and disease-free survival (e.g. no recurrence or metastasis occurred), expressed as adjusted hazard ratio with 95% confidence intervals and p values, from multivariate Cox regression analysis.

SECONDARY OUTCOMES:
5 year disease free survival between short and long time to treatment | 5 years after treatment
  5 year cumulative probability of disease free survival in patients with a short (<30 days) versus long (30 days or more) time to treatment, presented as percentages with 95% confidence intervals and p-values using Kaplan Meier survival curves and the log-rank test.
5 year disease specific survival between short and long time to treatment | 5 years after treatment
  5 year cumulative probability of disease specific survival in patients with a short (<30 days) versus long (30 days or more) time to treatment, presented as percentages with 95% confidence intervals and p-values using Kaplan Meier survival curves and the log-rank test.
5 year overall survival between short and long time to treatment | 5 years after treatment
  5 year cumulative probability of overall survival in patients with a short (<30 days) versus long (30 days or more) time to treatment, presented as percentages with 95% confidence intervals and p-values using Kaplan Meier survival curves and the log-rank test.
5 year disease free survival between participating centers | 5 years after treatment
  5 year cumulative probability of disease free survival in patients treated at the Maastricht University Medical Center+ versus Radboud University Medical Center, presented as percentages with 95% confidence intervals and p-values using Kaplan Meier survival curves and the log-rank test.
5 year disease specific survival between participating centers | 5 years after treatment
  5 year cumulative probability of disease specific survival in patients treated at the Maastricht University Medical Center+ versus Radboud University Medical Center, presented as percentages with 95% confidence intervals and p-values using Kaplan Meier survival curves and the log-rank test.
5 year overall survival between participating centers | 5 years after treatment
  5 year cumulative probability of overall survival in patients treated at the Maastricht University Medical Center+ versus Radboud University Medical Center, presented as percentages with 95% confidence intervals and p-values using Kaplan Meier survival curves and the log-rank test.

CONTACTS AND LOCATIONS:
Overall Officials: N Kelleners-Smeets, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (2):
- Netherlands (2):
  - Maastricht University Medical Center+, Maastricht
  - Radboud University Medical Center, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fania L, Didona D, Di Pietro FR, Verkhovskaia S, Morese R, Paolino G, Donati M, Ricci F, Coco V, Ricci F, Candi E, Abeni D, Dellambra E. Cutaneous Squamous Cell Carcinoma: From Pathophysiology to Novel Therapeutic Approaches. Biomedicines. 2021 Feb 9;9(2):171. doi: 10.3390/biomedicines9020171. PMID 33572373
- [Background] Kallini JR, Hamed N, Khachemoune A. Squamous cell carcinoma of the skin: epidemiology, classification, management, and novel trends. Int J Dermatol. 2015 Feb;54(2):130-40. doi: 10.1111/ijd.12553. Epub 2014 Nov 27. PMID 25428226
- [Background] Que SKT, Zwald FO, Schmults CD. Cutaneous squamous cell carcinoma: Incidence, risk factors, diagnosis, and staging. J Am Acad Dermatol. 2018 Feb;78(2):237-247. doi: 10.1016/j.jaad.2017.08.059. PMID 29332704
- [Background] Stern RS; PUVA Follow-Up Study. The risk of squamous cell and basal cell cancer associated with psoralen and ultraviolet A therapy: a 30-year prospective study. J Am Acad Dermatol. 2012 Apr;66(4):553-62. doi: 10.1016/j.jaad.2011.04.004. Epub 2012 Jan 20. PMID 22264671
- [Background] Stratigos AJ, Garbe C, Dessinioti C, Lebbe C, Bataille V, Bastholt L, Dreno B, Fargnoli MC, Forsea AM, Frenard C, Harwood CAlpha, Hauschild A, Hoeller C, Kandolf-Sekulovic L, Kaufmann R, Kelleners-Smeets NW, Malvehy J, Del Marmol V, Middleton MR, Moreno-Ramirez D, Pellecani G, Peris K, Saiag P, van den Beuken-van Everdingen MHJ, Vieira R, Zalaudek I, Eggermont AMM, Grob JJ; European Dermatology Forum (EDF), the European Association of Dermato-Oncology (EADO) and the European Organization for Research and Treatment of Cancer (EORTC). European interdisciplinary guideline on invasive squamous cell carcinoma of the skin: Part 1. epidemiology, diagnostics and prevention. Eur J Cancer. 2020 Mar;128:60-82. doi: 10.1016/j.ejca.2020.01.007. Epub 2020 Feb 26. PMID 32113941
- [Background] Phung D, Ahmadi N, Gupta R, Clark JR, Wykes J, Ch'ng S, Elliott MS, Palme CE, Shannon K, Wu R, Lee JH, Low TH. Survival outcomes of perineural spread in head and neck cutaneous squamous cell carcinoma. ANZ J Surg. 2022 Sep;92(9):2299-2304. doi: 10.1111/ans.17908. Epub 2022 Jul 22. PMID 35866314
- [Background] Brantsch KD, Meisner C, Schonfisch B, Trilling B, Wehner-Caroli J, Rocken M, Breuninger H. Analysis of risk factors determining prognosis of cutaneous squamous-cell carcinoma: a prospective study. Lancet Oncol. 2008 Aug;9(8):713-20. doi: 10.1016/S1470-2045(08)70178-5. Epub 2008 Jul 9. PMID 18617440
- [Background] Brougham ND, Dennett ER, Cameron R, Tan ST. The incidence of metastasis from cutaneous squamous cell carcinoma and the impact of its risk factors. J Surg Oncol. 2012 Dec;106(7):811-5. doi: 10.1002/jso.23155. Epub 2012 May 16. PMID 22592943
- [Background] Mourouzis C, Boynton A, Grant J, Umar T, Wilson A, Macpheson D, Pratt C. Cutaneous head and neck SCCs and risk of nodal metastasis - UK experience. J Craniomaxillofac Surg. 2009 Dec;37(8):443-7. doi: 10.1016/j.jcms.2009.07.007. Epub 2009 Aug 27. PMID 19713116
- [Background] Schmults CD, Karia PS, Carter JB, Han J, Qureshi AA. Factors predictive of recurrence and death from cutaneous squamous cell carcinoma: a 10-year, single-institution cohort study. JAMA Dermatol. 2013 May;149(5):541-7. doi: 10.1001/jamadermatol.2013.2139. PMID 23677079
- [Background] Kyrgidis A, Tzellos TG, Kechagias N, Patrikidou A, Xirou P, Kitikidou K, Bourlidou E, Vahtsevanos K, Antoniades K. Cutaneous squamous cell carcinoma (SCC) of the head and neck: risk factors of overall and recurrence-free survival. Eur J Cancer. 2010 Jun;46(9):1563-72. doi: 10.1016/j.ejca.2010.02.046. Epub 2010 Mar 24. PMID 20338745
- [Background] Peat B, Insull P, Ayers R. Risk stratification for metastasis from cutaneous squamous cell carcinoma of the head and neck. ANZ J Surg. 2012 Apr;82(4):230-3. doi: 10.1111/j.1445-2197.2011.05994.x. Epub 2012 Jan 31. PMID 22510179
- [Background] Yung AE, Crouch G, Varey AHR, Lo S, Elliott MS, Lee J, Rawson R, Gupta R, Hong AM, Clark JR, Ch'ng S. Benchmarking Survival Outcomes Following Surgical Management of pT3 and pT4 Cutaneous Squamous Cell Carcinoma of the Head and Neck. Ann Surg Oncol. 2022 Aug;29(8):5124-5138. doi: 10.1245/s10434-022-11669-z. Epub 2022 Apr 13. PMID 35419758
- [Background] van Hoeve JC, Vernooij RWM, Fiander M, Nieboer P, Siesling S, Rotter T. Effects of oncological care pathways in primary and secondary care on patient, professional and health systems outcomes: a systematic review and meta-analysis. Syst Rev. 2020 Oct 25;9(1):246. doi: 10.1186/s13643-020-01498-0. PMID 33100227
- [Background] Schutte HW, van den Broek GB, Steens SCA, Hermens RPMG, Honings J, Marres HAM, Merkx MAW, Weijs WLJ, Arens AIJ, van Engen-van Grunsven ACH, van Herpen CML, Kaanders JHAM, van den Hoogen FJA, Takes RP. Impact of optimizing diagnostic workup and reducing the time to treatment in head and neck cancer. Cancer. 2020 Sep 1;126(17):3982-3990. doi: 10.1002/cncr.33037. Epub 2020 Jul 7. PMID 32634271
- [Background] Rowe DE, Carroll RJ, Day CL Jr. Prognostic factors for local recurrence, metastasis, and survival rates in squamous cell carcinoma of the skin, ear, and lip. Implications for treatment modality selection. J Am Acad Dermatol. 1992 Jun;26(6):976-90. doi: 10.1016/0190-9622(92)70144-5. PMID 1607418
- [Background] Endo Y, Tanioka M, Miyachi Y. Prognostic factors in cutaneous squamous cell carcinoma: is patient delay in hospital visit a predictor of survival? ISRN Dermatol. 2011;2011:285289. doi: 10.5402/2011/285289. Epub 2011 Nov 14. PMID 22363846
- [Background] DeGraaff LH, Platek AJ, Iovoli AJ, Wooten KE, Arshad H, Gupta V, McSpadden RP, Kuriakose MA, Hicks WL Jr, Platek ME, Singh AK. The effect of time between diagnosis and initiation of treatment on outcomes in patients with head and neck squamous cell carcinoma. Oral Oncol. 2019 Sep;96:148-152. doi: 10.1016/j.oraloncology.2019.07.021. Epub 2019 Jul 30. PMID 31422206
- [Background] Shang C, Feng L, Gu Y, Hong H, Hong L, Hou J. Impact of Multidisciplinary Team Management on the Survival Rate of Head and Neck Cancer Patients: A Cohort Study Meta-analysis. Front Oncol. 2021 Mar 8;11:630906. doi: 10.3389/fonc.2021.630906. eCollection 2021. PMID 33763367
- See also: Integral cancer center Netherlands; incidence rates on cutaneous squamous cell carcinomas — http://iknl.nl/kankersoorten/huidkanker/registratie/incidentie